CLINICAL TRIAL: NCT00590629
Title: Benefit of Elevation of HDL-C on Cardiovascular Outcomes in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: General Clinical Research Center (GCRC) (Unknown); Kos Pharmaceuticals (Industry)
Responsible Party: Donna Polk, CSMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HDL3954; GCRC: Grant #MO1-RR00425; NCT00192010 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2007-12

CONDITIONS: Coronary Artery Disease
Keywords: Women with and without CAD
MeSH Terms: conditions — Coronary Artery Disease | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Niaspan — 1500 mg Niaspan for 16 weeks

SUMMARY:
Several risk factors including high cholesterol contribute to heart disease. We know that lowering triglycerides and raising HDL (protective cholesterol) in men reduces the risk for heart disease. We expect that women will share this same benefit because the combination of high triglycerides and low HDL appears to be a more important risk for heart disease in women. Niacin reduces triglycerides and raises HDL. We also expect to see improvement in markers of inflammation and clot formation and blood vessel health, which we hypothesize should all confer a reduced risk of heart disease in women.

Women already taking lipid lowering statin will receive niacin therapy. We will measure blood lipid levels, markers of inflammation and clotting as well as a non-invasive measure of blood vessel reactivity. After 3 months of therapy we will repeat these measures.

ELIGIBILITY:
Inclusion Criteria:

* Stable women on statin therapy with LDL-C between 90-135mg/dl and triglycerides > 150mg/dl

Exclusion Criteria:

* History of MI, PTCA or surgery within previous 3 months

  * Currently on Niaspan and unwilling to withdraw Niaspan therapy or known intolerance to niacin
  * Active or known gall bladder disease
  * Pregnant or nursing women
  * Significant comorbidity that precludes participation
  * Significant liver disease, active alcoholism, or LFT >1.5x's ULN at screening
  * Diabetes or glucose > 126 mg/dl at screening
  * PI perceived inability to comply with protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CSMC, Los Angeles, California, United States